CLINICAL TRIAL: NCT04573439
Title: Children's Protein Requirements With Physical Activity: The ChiPP Study
Brief Title: Protein Requirements for Active Children
Acronym: ChiPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 261235
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Dietary Supplement: Dietary supplement: Protein intake Oral consumption of hourly experimental meals. Includes 4 meals containing a mixture of free amino acids, carbohydrates and fats from a protein-free formula mixture.
  The last 4 meals will contain labelled 13C phenylalanine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Dietary supplement: Protein intake — Oral consumption of hourly experimental meals. Includes 4 meals containing a mixture of free amino acids, carbohydrates and fats from a protein-free formula mixture.
  The last 4 meals will contain labelled 13C phenylalanine.

SUMMARY:
There is reason to believe the current dietary reference intakes for dietary protein for children are too low. Furthermore, children with high levels of physical activity and fitness may require a higher requirement. To better understand the protein requirements in minimally and highly physically fit and active children 8-10 y old, investigators will use the indicator amino acid oxidation technique.

DETAILED DESCRIPTION:
Purpose: Determine dietary protein requirements using the indicator amino acid oxidation (IAAO) method in a group of thoroughly phenotyped school-age children who engage in different levels of Physical Activity.

Hypothesis: Daily dietary protein requirements are greater in children with high level of physical activity vs. sedentary children.

Justification: Adequate dietary protein intake is essential to support cellular integrity, physical growth and function. Although dietary protein malnutrition is not prevalent in the U.S., highly active individuals may require greater than the average protein intake to support both increased metabolic demands and skeletal muscle repair and remodeling. The current Institute of Medicine (IOM) guidelines do not have separate dietary protein estimated average requirement (EARs) for physically active children.

Research Design: This is a comparative two-group (sedentary vs. physically active), single center, prospective cohort study designed to estimate and compare the dietary protein requirements among sedentary and active children between the ages of 8-10 years. Each participant will be assigned to 7 one-day dietary protein levels with the goal of obtaining measures of phenylalanine oxidation corresponding to each level of protein intake.

Up to 30 children will be recruited for this study at the Arkansas Children's Nutrition Center (ACNC) with the expectation of a 20% attrition rate resulting in a total of 24 children (n=12/group) in the final analysis. The recruitment will ensure equal representation of both sexes of children. After screening, the children and parents will attend an in-person or remote assent/consent visit.

After the assent/consent visit, children will consume a 2-day run-in diet to ensure protein intakes of 1.5 g/kg/day and energy intakes of 1.7 x resting energy expenditure. Each child will participate in 7 testing days, following an overnight fast before each visit. At each of these testing days, participants will be randomly assigned to one of 7 test protein dosages (0.2-2.4 g·kg-1·d-1) consisting of 8 isocaloric and isonitrogenous meals provided hourly, each meal presenting 1/12 of the daily energy requirement. Study day diet is composed of a crystalline amino acid mixture based on the amino acid profile of egg protein and protein free diet toddler and 2 formulas for carbohydrate and fat. A stable isotope tracer will be added to the 5th through 8th meals. Investigators will measure the rate of oxidation of this tracer expired in breath (F13CO2), and flux of this tracer by its enrichment in urine.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  * Boys or girls
  * Ages 8-10 years
  * All races
  * All ethnicities
  * Children who were determined to have normal weight (BMI <85th percentile) already determined under Mitochondria (MI) Energy (IRB Protocol: 260376)
  * Participants willing to stop taking nutritional supplements (e.g., multivitamins, vitamin D, fish oil, probiotics, prebiotics, immune boosters, and others) for at least 2 weeks prior to each study testing visit
  * Children without an infection requiring antibiotics willing to be rescheduled after at least 2 months of finalizing antibiotic treatment.
  * Children without viral infections such as diarrhea, cold, or flu willing to be rescheduled after at least 2 weeks of resolution of symptoms.
  * Children determined sedentary or active, based on both peak oxygen uptake (VO2) and accelerometer data, as described below: Children who completed a peak fitness test during MI Energy (IRB Protocol: 260376), and for whom peak VO2 data are as follows:

Peak ⩒O2, ml·min-1·fat free mass index (FFMI)-1 Boys Girls Boys Girls

* 89 ≤ 80 ≥115 ≥105 FFMI, fat-free mass index

AND

Children who completed accelerometer measures during MI Energy (IRB Protocol: 260376), and for whom average daily activity counts and/or minutes of moderate to vigorous physical activity are as follow:

Sedentary Active Activity counts/day <2,924,494 ≥3,767,075 Minutes of Moderate to vigorous physical activity/day <60 ≥60

Children who completed National Survey of Children's Health and Youth Risk Behavior Survey (NSCH-YRBS) questionnaire during MI Energy study (IRB Protocol: 260376). Children who report ≥3 hours/day of Television (TV) (Sedentary) or ≤2 hours/day of TV (Active) will be considered

* Children who completed Dual-energy x-ray absorptiometry (DXA) measures during MI Energy study (IRB Protocol: 260376)
* Children whose parents consented to the following in the MI Energy study (IRB Protocol: 260376): o A) be contacted about future follow-up studies to MI Energy, and having the data that is collected about their child in MI Energy being used also in these follow-up studies; and

  * B) information collected in the MI Energy study may be used in future research related to bioenergetics (for example, blood cell mitochondria function), nutrition, obesity, cardiovascular health, or development; and
  * C) any biological samples collected in the MI Energy study may be used in future research related to bioenergetics (for example, blood cell mitochondria function), nutrition, obesity, cardiovascular health, or development.

Exclusion Criteria:

* • Participants who have been excluded from participation in the study MI Energy (IRB Protocol: 260376)

  * Participants whose parents report any change in medical history that may potentially affect participation and/or study outcomes as determined by PI
  * Weight loss >3 kg in last 6 months
  * Taking medications that knowingly influences protein metabolism
  * Phenylketonuria

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
13C Phenylalanine Oxidation | 8 hours
  Urine and breath will be collected during the study to measure the rate of 13C phenylalanine oxidation

CONTACTS AND LOCATIONS:
Overall Officials: Eva C Diaz Fuentes, MD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No